CLINICAL TRIAL: NCT03787368
Title: An Observer-blind, Multi-center, Placebo-controlled, Parallel Group Study to Assess the Safety and Tolerability and to Characterize the Pharmacokinetics and the Pharmacodynamics of Different Doses of BAY1213790 in Patients With End-stage Renal Disease Undergoing Hemodialysis
Brief Title: End-stage Renal Disease (ESRD) Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20046; 2018-003109-24 (EudraCT Number)
Record Dates: First submitted 2018-12-24; First posted 2018-12-26 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Renal Dialysis
Keywords: End-stage renal disease patients undergoing hemodialysis
MeSH Terms: interventions — osocimab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients, investigators, and all other site staff will remain blinded for the administered BAY1213790 or placebo, with the exception of the unblinded pharmacist or specifically dedicated site personnel.The sponsor will be not be blinded. Bioanalysis of plasma concentrations and PD parameters, as well as the evaluation of results will be performed in a non-blinded fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose 1 of BAY1213790 (Experimental): Single intravenous infusion BAY1213790 (Dose 1)
  Interventions: Drug: BAY1213790
- Dose 2 of BAY1213790 (Experimental): Single intravenous infusion BAY1213790 (Dose 2)
  Interventions: Drug: BAY1213790
- Placebo (Placebo Comparator): Single intravenous infusion placebo
  Interventions: Drug: 0.9% sodium chloride solution

INTERVENTIONS:
Drug: BAY1213790 — Single intravenous infusion of BAY1213790 (Two different doses)
  Arms: Dose 1 of BAY1213790; Dose 2 of BAY1213790
Drug: 0.9% sodium chloride solution — Single intravenous infusion of Placebo (0.9% sodium chloride solution)
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety of two different doses of a drug called BAY1213790 and how well it is tolerated in patients with end-stage renal disease (ESRD) undergoing hemodialysis (HD). Approximately 40, with up to 60 study patients will take part in the study.

ELIGIBILITY:
Inclusion Criteria

* Male and female patients between 18 and 80 years of age.
* ESRD on hemodialysis (including hemodiafiltration) for at least 3 months
* Life expectancy of > 6 months
* Women of non-childbearing potential

Exclusion Criteria:

* High risk for clinically significant bleeding
* Acute renal failure
* Planned major surgery in the next 7 months from randomization
* Concomitant use of oral anticoagulant therapy or antiplatelet therapy
* Documented thrombotic event in the past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Number of major and CRNM bleeding events | Approx. 4 weeks (Before study drug or placebo administration)
  CRNM bleeding: Clinically Relevant Non-Major bleeding
Number of major and CRNM bleeding events | Approx. 4 weeks (After study drug or placebo administration)

SECONDARY OUTCOMES:
AUC (AUC(0-tlast) will be used as main parameter if mean AUC(tlast-∞) >20% of AUC) | Approx. 5 months (Pre-dose to follow up)
  AUC: Area under the concentration vs. time curve from zero to infinity after single (first) dose
aPTT will be measured via the kaolin-trigger method (clotting assay) | Approx. 6 months (Before study drug or placebo administration to follow up)
  aPTT: activated Partial Thromboplastin Time
Factor XI activity will be assessed with an aPTT-based coagulation test using FXI | Approx. 6 months (Before study drug or placebo administration to follow up)
  FXI: Factor XI

CONTACTS AND LOCATIONS:
Locations (15):
- United States (4):
  - California Institute of Renal Research - Chula Vista, Chula Vista, California
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Research by Design, LLC, Chicago, Illinois
  - Renal and Transplant Associates of New England, PC, Springfield, Massachusetts
- Belgium (3):
  - CHU de Charleroi Hôpital civil, Lodelinsart, Hainaut
  - UZ Brussel, Bruxelles - Brussel
  - UZ Leuven Gasthuisberg, Leuven
- Portugal (3):
  - CHLO - Hospital Santa Cruz, Carnaxide, Lisbon District
  - Pluribus Dialise - Cascais (DaVita), Cascais, Lisbon District
  - CHMT - Hospital Rainha Santa Isabel, Torres Novas, Santarém District
- Spain (5):
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Ciutat Sanitària i Universitària de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.